CLINICAL TRIAL: NCT05156931
Title: Exploration of Patient Self-medication Practices During and After Cancer in France: Cross-sectional Observational Study With Online Response
Brief Title: Exploration of Patient Self-medication Practices During and After Cancer in France
Acronym: CASEME
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 BALAYSSAC
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2021-12

CONDITIONS: Cancer; Self-medication
Keywords: cancer; self-medication; quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the patient self-medication practices during and after cancer in France, using an online questionnaire

DETAILED DESCRIPTION:
Patients will be contacted by email from patient's associations. Patients will be informed of the objectives of the study and will be free to answer or not to the online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Past or active cancer

Exclusion Criteria:

* Speaking French
* Not living in France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients contacted by cancer patient's association
Sampling Method: Non-Probability Sample
Enrollment: 681 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Self-medication | day 1
  declaration of a practice of self-medication

SECONDARY OUTCOMES:
Class of products used in self-medication | day 1
  non-prescription medicine, herbal medicine, aromatherapy, homeopathy, and food supplements
Indication for self-medication | day 1
  For treatment of side-effects, improvements in anti-cancer effects
Origin of self-medication products | day 1
  pharmacy, market, internet, other
Perception of adverse effects and drug-drug interaction related to self medication | day 1
  yes / no
QLQ-C30 questionnaire | day 1
  Global health status Functional scales Physical functioning Role functioning Emotional functioning Cognitive functioning Social functioning Fatigue Nausea and vomiting Pain Dyspnoea Insomnia Appetite loss Constipation Diarrhoea Financial difficulties

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No